CLINICAL TRIAL: NCT04882709
Title: Using Headphone Presentation to Investigate Compression Strategy Modifications in Hearing Aids for Moderate-to-severe Hearing Loss
Brief Title: Compression Headphone Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No reliable differences across conditions, unacceptable test-retest reliability
Sponsor: Sonova AG (Industry)
Collaborators: Sonova Canada Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 365
Record Dates: First submitted 2021-05-04; First posted 2021-05-12 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The acoustic output of the different devices had been recorded and the recordings have been presented in random order (random order created by the sound survey algorithm) to the participants in a digital sound survey, so neither the researcher nor the participant knew which recording the participant was listening to when rating.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Hearing aid 1 default amplification strategy (Experimental): Hearing aid 1 default amplification strategy: A receiver-in-canal (RIC) hearing aid developed by the study sponsor used with the default settings as specified in the study sponsor's fitting software.
  Interventions: Device: Recording with hearing aid
- Hearing aid 2 (Experimental): Hearing aid 2: A receiver-in-canal (RIC) hearing aid developed by the another hearing aid manufacturer used with the default settings as specified in the manufacturer's fitting software.
  Interventions: Device: Recording with hearing aid
- Hearing aid 1 strategy 1 (Experimental): Hearing aid 1 strategy 1: A receiver-in-canal (RIC) hearing aid developed by the study sponsor used with a modified compression strategy that is expected to improve sound quality.
  Interventions: Device: Recording with hearing aid
- Hearing aid 1 strategy 2 (Experimental): Hearing aid 1 strategy 2: A receiver-in-canal (RIC) hearing aid developed by the study sponsor used with a modified compression strategy that is expected to improve sound quality.
  Interventions: Device: Recording with hearing aid
- unaided (No Intervention): Unaided recording to be used for normalization of rating results.

INTERVENTIONS:
Device: Recording with hearing aid — Each participant will listen to sound samples via headphones. Sound samples have been recorded with a hearing aid that was set to each participant's individual hearing loss and different amplification strategies, and an unaided reference. Participants will be asked to rate different aspects of sound quality while listening to the different sound samples.
  Arms: Hearing aid 1 default amplification strategy; Hearing aid 1 strategy 1; Hearing aid 1 strategy 2; Hearing aid 2

SUMMARY:
The stimuli consist of speech in quiet, speech in noise, reverberant speech, and music recorded with different hearing aid settings, post-processed for headphone presentation and incorporated in an online sound survey. Participants will receive tablets and headphones to conduct a sound quality rating at home. The survey will involve a training session and within-subject repeated measures. Stimuli presentation will be randomized by sound quality rating tool.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-99 years) with ≥3 months hearing aid experience
* binaural, symmetric, sensorineural N3 to N4 hearing loss
* able to use Android interface and receive a video call on phone/computer
* fluent in English

Exclusion Criteria:

* children/teenagers
* normal hearing or hearing loss exceeding N4 by 10dB
* cannot wear over-ear headphones

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinyu Qian, PhD, Principal Investigator — Sonova Canada Inc.
Locations (1):
- Sonova Innovation Centre Toronto, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sound Survey: Each participant will conduct a sound survey at home with equipment (tablet and headphones) that were shipped to the participant's place of residence. During the survey, sound samples were randomly assigned to the push buttons participants were clicking to listen to a sound:
  Hearing aid 1 default amplification strategy: A receiver-in-canal (RIC) hearing aid developed by the study sponsor used with the default settings as specified in the study sponsor's fitting software.
  Hearing aid 2: A receiver-in-canal (RIC) hearing aid developed by the another hearing aid manufacturer used with the default settings as specified in the manufacturer's fitting software.
  Hearing aid 1 strategy 1: A receiver-in-canal (RIC) hearing aid developed by the study sponsor used with a modified compression strategy that is expected to improve sound quality.
  Hearing aid 1 strategy 2: A receiver-in-canal (RIC) hearing aid developed by the study sponsor used with a modified compression strategy that is expected to improve sound quality.
  Unaided: Recordings made without hearing aids. Ratings for this sound sample were used for normalization of survey results.
Period: Overall Study
Arm/Group | Sound Survey
Started | 12 (Randomization was assigned automatically for each trial and the researchers were blinded to how many participants listened to a specific condition first.)
Hearing Aid 1 Default Amplification Strategy | 12
Hearing Aid 2 | 12
Hearing Aid 1 Strategy 1 | 12
Hearing Aid 1 Strategy 2 | 12
Unaided | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Collected data was based on self-reports or data provided by the participants, and available information in our participant database. One successfully completed study participant's data set, which was collected in the early phase of the study design, was excluded from the analysis because the stimuli were changed afterwards. The analysis does not contain any of this participant's data or information, bringing the total number of analyzed participants down to 11.
Groups:
- Complete Sample: Each participant will listen to sound samples via headphones. Sound samples have been recorded with each of the devices listed under "intervention" which were set to each participant's individual hearing loss, and an unaided reference. Participants will be asked to rate different aspects of sound quality while listening to the different sound samples.
Arm/Group | Complete Sample
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hearing aid experience [Mean (Standard Deviation); unit: years] | 17 (10)
Hearing loss [Count of Participants; unit: Participants] | 11
Normal or corrected to normal vision [Count of Participants; unit: Participants] | 11
Good cognitive abilities [Count of Participants; unit: Participants] | 11

OUTCOME MEASURES:

1. Primary Outcome: Sound Quality Rating
Description: Participants moved through a self-guided, double-blinded sound survey which presented sound samples of all hearing aid conditions (see Arms/Groups for conditions) and asked participants to rate the sound quality dimensions on a scale. The rating dimensions and scales were based on a sound quality rating guidance document by Delta Labs (Danmark) ranging from 0 to 100 with step sizes of 1 and descriptive markers at 0 (worst), 20, 40, 60, 80 and 100 (best) depending on the dimension (Reverberation (only assessed for Speech in Quiet and Reverberant Speech), Sound Source Localization, Sound Source Separation, and Timbral Balance). Overall Preference was implemented as a ranking according to the 5-point Mean Opinion Score (bad (1), poor (2), fair (3), good (4), excellent (5); MOS, International Telecommunication Union, 1996).
Time Frame: 1 hour
Population: The median and IQR is presented for each sound quality dimension (Reverberation, Sound Source Separation, Sound Source Location and Overall) in sound scene (speech in quiet, speech in noise, speech in reverberance, music).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Hearing Aid 1 Default Amplification Strategy: A receiver-in-canal (RIC) hearing aid developed by the study sponsor used with the default settings as specified in the study sponsor's fitting software.
- Hearing Aid 2: A receiver-in-canal (RIC) hearing aid developed by the another hearing aid manufacturer used with the default settings as specified in the manufacturer's fitting software.
- Hearing Aid 1 Strategy 1; Hearing Aid 1 Strategy 2: A receiver-in-canal (RIC) hearing aid developed by the study sponsor used with a modified compression strategy that is expected to improve sound quality.
- Unaided: A recording without any amplification.
Arm/Group | Hearing Aid 1 Default Amplification Strategy | Hearing Aid 2 | Hearing Aid 1 Strategy 1 | Hearing Aid 1 Strategy 2 | Unaided
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
units on a scale
  Reverberation in speech in quiet | 69 [55 to 75] | 55 [28.75 to 70.75] | 71 [64.75 to 87.75] | 80 [47.5 to 90] | 42 [26 to 59]
  Reverberation in reverberant speech | 56.5 [50.25 to 72] | 54.5 [41 to 70.5] | 70 [60.75 to 80.75] | 70.5 [51.25 to 73.75] | 40.5 [21 to 55.25]
  Sound source location in speech in quiet | 59 [54.25 to 70.75] | 50.5 [39.5 to 67] | 61.5 [52.75 to 78] | 55 [51.25 to 61.5] | 25 [16 to 37.5]
  Sound source location in speech in noise | 74 [63 to 80.25] | 63 [44.75 to 73] | 65 [50 to 78.5] | 61 [57.75 to 76.75] | 43.5 [25.5 to 62.75]
  Sound source localization in reverberant speech | 45.5 [36.25 to 60.5] | 56 [41.5 to 63] | 69.5 [51 to 73] | 55.5 [50.75 to 67.25] | 49 [30.75 to 59.5]
  Sound source localization in music | 60.5 [53 to 66.25] | 69.5 [60.25 to 74] | 66.5 [63 to 71] | 67.5 [59.75 to 78.75] | 44 [24.25 to 56.25]
  Sound source separation in speech in quiet | 62.5 [53.25 to 74] | 59 [56.75 to 71.25] | 59.5 [55.75 to 74] | 69 [52 to 76.75] | 29 [16.5 to 41.25]
  Sound source separation in speech in noise | 55 [46.75 to 57.25] | 52 [40 to 60.25] | 70 [53.5 to 75.25] | 64.5 [50.75 to 69] | 30 [16 to 40]
  Sound source separation in reverberant speech | 50 [36.75 to 54.5] | 61 [39.5 to 76] | 61 [53.25 to 65.25] | 61 [47.5 to 70.75] | 39 [30.25 to 55.5]
  Sound source separation in music | 65.5 [51.5 to 79.25] | 71.5 [40 to 76.75] | 68.5 [53 to 77.25] | 79.5 [71 to 80.5] | 30 [15.75 to 61.75]
  Overall Preference for speech in quiet | 3.5 [2.5 to 4] | 3.5 [3 to 3.5] | 3.5 [3.5 to 4] | 4 [3.25 to 4] | 1 [1 to 1]
  Overall Preference for speech in noise | 3.5 [3.5 to 4] | 3.5 [2.25 to 4] | 3.5 [3 to 3.75] | 3 [3 to 3.75] | 1 [1 to 3]
  Overall Preference for reverberant speech | 3 [1.75 to 3.5] | 3 [2 to 4] | 4 [3.5 to 4] | 3.5 [3 to 4] | 3 [1.25 to 3.5]
  Overall Preference for music | 3 [2.25 to 3.75] | 3 [2.75 to 4.5] | 3.5 [3 to 3.75] | 4 [3.5 to 4] | 1 [1 to 3]

ADVERSE EVENTS:
Time Frame: Data were collected as long as a participant was enrolled in the study, which was from the first to the second appointment. This time frame was about 2 weeks for each participant.
Description: Point of Care Risk Assessment conducted at each visit, including questions regarding overall health.
Groups:
- Complete Sample: Each participant will conduct a sound survey at home with equipment (tablet and headphones) that were shipped to the participant's place of residence.
Arm/Group | Complete Sample
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT04882709/Prot_SAP_000.pdf